CLINICAL TRIAL: NCT01311934
Title: Clinical Application of the Spectrum of Visceral Stiffness Measurement Using Acoustic Radiation Force Impulse Technology
Brief Title: Visceral Stiffness Measurement Using Acoustic Radiation Force Impulse
Acronym: ARFI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sheng-Hung Chen, China Medical University Hospital
Other Study IDs: DMR100-IRB-001
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Visceral Stiffness; Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HBV-infected
- HCV-infected

SUMMARY:
The acoustic radiation force impulse (ARFI) technology provides real-time measurements of tissue stiffness.

Aim: Using the ARFI ultrasonography, the investigators aims are to complete the correlation and validity studies between visceral ARFI quantification and the referenced Metavir fibrosis scoring and to conduct subsequent innovative studies on liver diseases.

DETAILED DESCRIPTION:
Using ARFI technology, we are establishing a complete hepatic and visceral shear wave spectrum to correspond to the entire METAVIR fibrosis scoring and various functional stratifications.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic liver diseases who underwent liver biopsy
* patients with pathologically or radiologically proven cirrhosis

Exclusion Criteria:

* Post major abdominal surgery
* After interferon or neucleos(t)ides treatment
* PBC,PSC,WD,AIH,viral coinfections
* Liver abscess
* Exposure to hepatotoxic drugs or chemicals
* Thrombosis of splenic vein, portal veins
* After resection or embolism of the spleen
* Acute or chronic pancreatitis
* Biopsy contraindications (not exclusive)
* ARFI measurements low quality
* Fibrotest contraindications:

Acute hepatitides, Extrahepatic cholestasis, e.g., pancreatic cancer, gallstones, CBD>0.7cm Severe hemolysis

* Cardiac congestion
* Liver cancer other than HCC
* Treated HCC

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver diseases
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hung Chen, MD, Principal Investigator — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital; Cheng-Yuan Peng, MD,PhD, Study Director — Hepatogastroenterology, Department of Internal Medicine, China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan